CLINICAL TRIAL: NCT05711732
Title: Collection of Plasma Samples Using Sodium Heparin From Subjects Undergoing Intravenous Busulfan Treatment
Brief Title: Busulfan Sample Collection Study
Status: Recruiting | Type: Observational
Sponsor: Saladax Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SBI-BSF-001
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Subjects Treated With Busulfan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: MyCare Oncology Busulfan Assay Kit — This is a sample collection study only. Patient treatment will not be determined by the outcome of the analytical test results.

SUMMARY:
Busulfan (Busulfex®) is an alkylating drug used as a conditioning regimen prior to allogeneic hematopoietic stem cell transplantation. Busulfan has wide inter- and intra-patient pharmacokinetic variability resulting in variable exposure leading to increased risk of toxicities or sub-optimal treatment outcomes. Therapeutic drug monitoring of busulfan using patient plasma samples would benefit clinicians by providing the ability to personalize the dose to achieve a target busulfan exposure.

DETAILED DESCRIPTION:
This protocol is sponsored by Saladax Biomedical, Inc (SBI). The protocol involves the use of sodium heparin plasma sample collected from human subjects receiving intravenous busulfan treatment for the use in the development of a diagnostic test for this drug. A subset of 10 enrolled subject samples will be tested on site using an automated immunoassay MyCareTM Oncology Busulfan Assay Kit manufactured by SBI.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric and adult female or male subjects;
2. Current treatment with intravenous busulfan with documentation of diagnosed malignant hematologic or non-malignant disease condition requiring treatment;
3. Adult participants must be capable of understanding and providing written informed consent, approved by an Institutional Review Board (IRB) prior to the initiation of any screening or study-specific procedures. Participants less than 18 years old must provide written assent with appropriate consent provided by legal guardian, who must be capable of understanding and providing informed consent, per Institutional Review Board (IRB) procedures, prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

1. Unwilling or unable to follow protocol requirements or to give written informed consent;
2. Patients receiving oral busulfan (e.g., Myleran®) treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 150 unique subjects across participating sites consisting of males and females who meet the protocol Inclusion/ Exclusion criteria as described above. Multiple (3 to 12) plasma samples by venous draw will be collected from each subject for a single day of busulfan dosing. Sample collection timing used to inform dose calculation shall be performed per the site standard of clinical care for patients prescribed busulfan.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Method Comparison Study | Sample collection to take place over 1 year. Samples to be analyzed monthly.
  The samples being collected according to the protocol, SBI-BSI-001, will be used to compare the quantitate determination of BSF in patient samples based on the immunoassay vs. LC-MS/MS methods .

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - The University of Texas MD Anderson Cancer Center, Houston, Texas